CLINICAL TRIAL: NCT00279656
Title: Collaborative Approach to Improve the Quality of Medicines Use in Elderly Inpatients - Randomized Controlled Trial
Brief Title: Benefit of a Collaborative Approach to Improve the Quality of Medicines Use in Elderly Inpatients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: om050-40/2003
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2006-01-19 (Estimated); Status verified 2004-06

CONDITIONS: Frail Elderly Inpatient
Keywords: Frail elderly; Pharmaceutical services; Drug therapy; Geriatrics; Randomized controlled trial; Hospitals, teaching
MeSH Terms: interventions — Pharmaceutical Services

INTERVENTIONS:
Behavioral: Pharmaceutical care

SUMMARY:
The purpose of this study is to evaluate the impact of a collaborative approach (geriatric care involving the collaboration with a clinical pharmacist) to optimize the prescription of medicines for elderly inpatients.

DETAILED DESCRIPTION:
Widespread evidence reveals frequent inadequate use of medicines in elderly patients. This includes inappropriate prescribing (overuse, underuse, misuse) that can lead to adverse drug events and drug-related admissions to hospital. In addition, when a patient is transferred from acute care settings to ambulatory care settings, discrepancies in medicines used often occur and can be hazardous.

Despite this, only limited data exist on the effectiveness of optimization strategies targeted at frail elderly inpatients.

Comparison: elderly inpatients receiving geriatric evaluation and management (GEM) care versus elderly inpatients receiving pharmaceutical care in addition to GEM care.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted on the acute geriatric unit of the university teaching hospital Mont-Godinne, Belgium

Exclusion Criteria:

* a terminal illness and life expectancy of less than 3 month
* expected length of stay of 2 days or less
* transfer from another unit where the patient had already been cared for by a GEM team
* refusal to participate
* inclusion during previous admission
* no time for the clinical pharmacist to compound the abstracted chart within 3 days of admission

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180
Dates: Start 2003-11; Study Completion 2005-06

PRIMARY OUTCOMES:
Appropriateness of prescribing (using the Medication Appropriateness Index, the Beers criteria, and the ACOVE criteria of underuse) on admission, at discharge, and 3 months post-discharge

SECONDARY OUTCOMES:
Polymedication on admission, at discharge, and 1,3,12 months after discharge
Mortality, readmission to hospital and visit to the emergency department 1,3,12 months after discharge
Satisfaction with information received on medicines

CONTACTS AND LOCATIONS:
Overall Officials: Anne Spinewine, MSc, Principal Investigator — Université Catholique de Louvain; Christian Swine, MD, Study Chair — Université Catholique de Louvain; Paul M Tulkens, PhD, Study Director — Université Catholique de Louvain
Locations (1):
- Université catholique de Louvain, Brussels, Belgium